CLINICAL TRIAL: NCT00018720
Title: Regulation of Sterol Homeostasis
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: GAST-026-95F
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-12

CONDITIONS: Hypertriglyceridemia
Keywords: triglyceride; bile acids; cholelithias
MeSH Terms: conditions — Hypertriglyceridemia

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to determine how people with high triglycerides metabolize and absorb bile acids, compounds made in the body from cholesterol.

This project has two objectives: A) To define the mechanism of impaired bile acid absorption in hypertriglyceridemia (specifically we will determine if the active or passive component of absorption is abnormal) and B) to determine the contribution of an alternative pathway of bile acid synthesis which begins with 27-hydroxylation of cholesterol. Because 27-hydroxylase is present in endothelial cells as well as liver, this pathway may play a role in removal of cholesterol from incipient atherosclerotic plaque.

ELIGIBILITY:
Hypertriglyceridemia and normal controls with normal lipids

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 1996-04; Study Completion 2000-12

CONTACTS AND LOCATIONS:
Overall Officials: Norman Javitt, M.D.; Alan Hofmann, M.D.; Loren Zech, M.D.
Locations (1):
- VA Medical Center, Minneapolis, Minnesota, United States